CLINICAL TRIAL: NCT03356067
Title: A Randomized, Sham and Cross-Over-Controlled Trial of Per-oral Endoscopic Pyloromyotomy (G-POEM) in Patients With Refractory Gastroparesis
Brief Title: Endoscopic Pyloromyotomy for Refractory Gastroparesis
Acronym: GREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); KU Leuven (Other); King's College Hospital NHS Trust (Other); University Hospital Augsburg (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Karolinska Institutet (Other); University of Amsterdam (Other); University Hospital Trnava (Network); Rigshospitalet, Denmark (Other); Comenius University (Other); Pavol Jozef Safarik University (Other); University of Chicago (Other); University of Cluj Napoca (Unknown); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Doc. (Ass. prof.) Jan Martinek, MD, PhD, AGAF, Ass. prof., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IClinicalEM2
Record Dates: First submitted 2017-10-27; First posted 2017-11-29 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Pyloromyotomy

STUDY DESIGN:
Intervention Model Description: Randomized sham-procedure controlled trial with crossover after 6 months after procedure
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esophago-gastro-duodenoscopy (Sham Comparator): Standard endoscopic examination of the upper GI tract with flexible endoscope.
  Interventions: Procedure: Esophago-gastro-duodenoscopy
- Gastric endoscopic peroral pyloromyotomy (Experimental): Experimental per-oral endoscopic myotomy of the pyloric sphincter
  Interventions: Procedure: Gastric endoscopic peroral pyloromyotomy

INTERVENTIONS:
Procedure: Gastric endoscopic peroral pyloromyotomy — G-POEM is, in principle, adaptation of POEM (per-oral endoscopic myotomy) in the stomach. The procedure consists of:
  1. Mucosal incision at the greater curvature 3-5 cm from the pylorus
  2. Submucosal tunnelling
  3. Finding pyloric sphincter
  4. Myotomy (2-3 cm) of the pyloric muscle
  5. Incision closure (endoclips or suture device)
  Other Names: G-POEM
  Arms: Gastric endoscopic peroral pyloromyotomy
Procedure: Esophago-gastro-duodenoscopy — Standard endoscopic examination of the upper GI tract with flexible endoscope
  Arms: Esophago-gastro-duodenoscopy

SUMMARY:
Gastroparesis is a disorder triggered by numerous causes and it is defined by symptoms and with an objective evidence of delayed gastric emptying in the absence of obstruction.

Effective treatment for gastroparesis is challenging especially in patients with severe symptoms. In refractory gastroparesis, endoscopic or surgical treatments may therefore be considered. Endoscopic treatments include intrapyloric injection of botulinum toxin and transpyloric insertion of a metallic stent. Surgical options involve implantation of a gastric "pacemaker" (gastric stimulation), pyloroplasty and subtotal gastrectomy.

Recently, a new endoscopic technique, gastric endoscopic per oral pyloromyotomy (G-POEM) has been introduced with promising preliminary results.

The aim of this prospective, sham-controlled, cross-over study (cross-over for patients randomized to the sham arm) is to compare short and long-term efficacy and safety of G-POEM in patients with refractory gastroparesis. Symptoms and objective parameters of gastric emptying will be the main outcome criteria. The reason of using a sham protocol is to control for the potential confounders (therapeutic effects of touch and belief, which are components of the placebo effect).

DETAILED DESCRIPTION:
Gastroparesis is a disorder triggered by numerous causes and it is defined by symptoms and with an objective evidence of delayed gastric emptying in the absence of obstruction (albeit pyloric spasms may play a role in a subset of patients). Gastroparesis may be a consequence of medication, surgery or diabetes but in approximately one third of patients, the cause remains unknown and the patients are diagnosed with idiopathic gastroparesis. Effective treatment for gastroparesis is challenging especially in patients with severe symptoms. The efficacy of prokinetics is dubious since they have not proven real clinical efficacy in placebo controlled trials. In refractory gastroparesis, endoscopic or surgical treatments may therefore be considered. Endoscopic treatments include intrapyloric injection of botulinum toxin and transpyloric insertion of a metallic stent. Surgical options involve implantation of a gastric "pacemaker" (gastric stimulation), pyloroplasty and subtotal gastrectomy. The partial effectiveness of botulinum toxin injection, stents and pyloroplasty suggests that disruption of the pyloric muscle may lead to a decreased intrapyloric tone and consequently to a symptomatic improvement in some patients with refractory gastroparesis.

Recently, a new endoscopic technique, gastric endoscopic per oral pyloromyotomy (G-POEM) has been introduced with promising preliminary results. Uncontrolled studies with so far limited number of patients have demonstrated a significant symptomatic improvement in approximately 70% of patients and improved or normalized of gastric emptying in more than a half of patients after G-POEM. A prospective uncontrolled study suggested that patients with idiopathic or post-surgical gastroparesis experiences higher success rate after G-POEM (70-80%) compared to patients with diabetic gastroparesis (50%).

G-POEM is, in principle, adaptation of POEM (per-oral endoscopic myotomy) in the stomach. POEM is now considered a standard treatment for esophageal achalasia and it has been shown to be safe and effective. In contrast to achalasia, pathophysiology of pyloric function in patients with gastroparesis is less understood and the explanation of how and why G-POEM should work is some-how hypothetical. For example, presumed pylorospasm has not been demonstrated as the predictive factor for treatment success of G-POEM yet. Refractory gastroparesis is often accompanied by psychological or even psychiatric disturbances and hence a placebo" effect of G-POEM cannot be ruled out. Therefore, the real clinical efficacy of G-POEM can only be demonstrated in a clinical randomized sham-controlled trial.

To assess the severity of gastroparesis-related symptoms, the Gastroparesis Cardinal Symptom Index (GCSI) has been developed for this item. The GCSI is part of a larger questionnaire PAGI-SYM (Patient Assessment of Upper Gastrointestinal Symptom severity index) established for assessment of patient-reported symptoms in gastroparesis (dyspepsia and gastroesophageal reflux). PAGI-SYM as well as GCSI subscale scores varied significantly by global disease severity, with higher (worse) scores observed in those subjects who rated their gastroparesis as moderate to severe.

The aim of this prospective, sham-controlled, cross-over study (cross-over for patients randomized to the sham arm) is to compare short and long-term efficacy and safety of G-POEM in patients with refractory gastroparesis. Symptoms and objective parameters of gastric emptying will be the main outcome criteria. The reason of using a sham protocol is to control for the potential confounders (therapeutic effects of touch and belief, which are components of the placebo effect).

Investigators plan to randomize 86 patients (43 in the active arm, ratio 1:1 active vs. sham). Sample size is calculated based on expected therapeutic success of G-POEM in 50% of patients vs. 20% in the sham group; significance level 0,05; study power 0,8; beta error 0,2; adjustment for 15% expected drop out.

Patients will be randomised in blocks of 6, stratified according to the etiologies: (idiopathic, diabetic, and post-surgical; patients after esophagectomy with gastric pull-through will not be included). Control visits will be scheduled at 3, 6, 12, 24, and 36 months. The primary outcome will be the proportion of patients with treatment success in the active group vs. sham group at 6 months after the procedure. Several secondary outcomes will also be assessed, including procedure-related parameters and safety parameters and change in Gastric Emptying Study (GET) after G-POEM vs. sham. After 6 months, patients randomized to the sham group will be offered G-POEM procedure and further followed up (cross-over part of the study) providing that they did not have a therapeutic effect of the sham procedure.

ELIGIBILITY:
Inclusion Criteria:

* Refractory (> 6 months) and severe (based on a validated total GSCI = Gastroparesis Cardinal Symptom Index) gastroparesis, with confirmed gastric emptying based on a gastric emptying study: standardized protocol of scintigraphy in all patients (performed less than 4 months prior to enrolment), or confirmed by a validated gastric emptying breath test [27]. The total GSCI score must be >2.3 [28].
* Abnormal gastric emptying is defined as retention of Tc-99 m >60% at 2 h and/or ≥10% of residual activity at 4 h on a standardized sulphur colloid solid-phase gastric emptying study.
* Radiolabelled liquids emptying study will be reserved as alternative technique for patients with poor tolerance of solids during scintigraphy. Abnormal gastric emptying will represent >50% retention of radiolabelled content (e.g. In-111) at 1 hour.
* Abnormal gastric empyting breath test based on a solid normal range determination for the test used (e.g. T1/2 > 109 min)

Exclusion Criteria:

* Age less than 18 years
* No previous attempt with at least one prokinetic drug
* No previous attempt to withdraw anticholinergic agents and glucagon like peptide -1 (GLP-1) and amylin analogues* in patients treated with these substances
* Active treatment with opioids or a history of treatment with opioids within 12 months before enrolment.
* Previous gastric surgery BI or II, esophagectomy, gastric pull-through
* Previous pyloromyotomy or pyloroplasty
* Known eosinophilic gastroenteritis
* Organic pyloric (or intestinal) obstruction (fibrotic stricture, etc.)
* Severe coagulopathy
* Esophageal or gastric varices and /or portal hypertensive gastropathy
* Advanced liver cirrhosis (Child B or Child C)
* Active peptic ulcer disease
* Pregnancy or puerperium
* Malignant or pre-malignant gastric diseases (dysplasia, gastric cancer, GIST)
* Any other condition, which in the opinion of the investigator would interfere with study requirements
* Uncontrolled diabetes mellitus
* Diagnosis of rumination syndrome or "eating" disorder (mental anorexia, bulimia nervosa) **
* Severe constipation without using laxatives
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Main outcome is the proportion of patients with treatment success after the procedure. | 6 months
  Treatment success is defined as a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score at least 50% from the baseline

SECONDARY OUTCOMES:
Proportion of patients with treatment success in the active arm after 3 months | 3 months
  Treatment success is defined as a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score at least 50% from the baseline
Proportion of patients with treatment success in the active arm after 12 months | 12 months
  Treatment success is defined as a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score at least 50% from the baseline
Proportion of patients with treatment success in the active arm after 24 months | 24 months
  Treatment success is defined as a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score at least 50% from the baseline
Proportion of patients with treatment success in the active arm after 36 months | 36 months
  Treatment success is defined as a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score at least 50% from the baseline
Proportion of patients with treatment success in the sham group at 3M | 3 months
  Treatment success is defined as a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score at least 50% from the baseline
Change in Gastroparesis Cardinal Symptom Index (GCSI) before and after G-POEM at 3, 6, 12, 24 and 36M and before vs. after sham procedure at 3M and 6M; | 3, 6, 12, 24 and 36 months
  Comparison of the change of the scores between the active and sham groups.
Change in The Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) before and after G-POEM at 3, 6, 12, 24 and 36M and before vs. after sham procedure at 3M and 6M; | 3, 6, 12, 24 and 36 months
  Comparison of the change of the scores between the active and sham groups.
Proportion of crossed-over patients with treatment success after 6 moths | 12 months
  Treatment success is defined as a decrease of a total GSCI symptom score at least 50% from the baseline
Change in Gastroparesis Cardinal Symptom Index (GCSI) crossed-over patients after the G-POEM procedure | 12 months
  Comparison of the change of the scores pre and post-procedure
Change in The Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) in crossed-over patients after the G-POEM procedure | 12 months
  Comparison of the change of the scores pre and post-procedure
Subgroup post-hoc analyses of the treatment success and change in symptomatic scores according to etiology of gastroparesis. | 3, 6, 12, 24 and 36 months
  Treatment success is defined as a decrease of a total GSCI symptom score at least 50%, change in GCSI and PAGY-SYM scores
Change in gastric emptying (scintigraphy) study and/or gastric emptying breath test before and after both G-POEM and sham procedure | 3, 6, 12, 24 and 36 months
  Comparison of the mean change of these parameters between active and sham groups.
Procedure details | 1 month
  length of the procedure
Procedural adverse events | 1 month
  perioperative adverse events (complications)
Long term adverse events | 3, 6, 12, 24 and 36 months
  Incidence rate of adverse events in treatment and sham groups

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, MD, PhD, Principal Investigator — University Medical Center Hamburg- Eppendorf | UKE Department for Interdisciplinary Endoscopy, Germany; Jan Martinek, MD, PhD, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic
Locations (14):
- University of Chicago, Chicago, Illinois, United States
- Belgium (2):
  - Department of Hepatogastroenterology at Cliniques universitaires St-Luc, Brussels, Belgium, Brussels
  - Translational Research in GastroIntestinal Disorders, Leuven, Belgium, Leuven
- Czechia (2):
  - Institute for Clinical and Experimental Medicine, Prague, Prague
  - University Hospital in Hradec Kralove, Hradec Králové
- The Department of Surgical Gastroenterology L, Denmark, Aarhus, Denmark
- Germany (2):
  - III. Medizinische Klinik, Medical Center/Klinikum Augsburg, Germany, Augsburg
  - University Medical Center Hamburg- Eppendorf | UKE Department for Interdisciplinary Endoscopy, Germany, Hamburg- Eppendorf
- Department of Gastroenterology and Hepatology, Amsterdam, The Netherlands, Amsterdam, Netherlands
- Regional Institute of Gastroenterology, Cluj-Napoca, Romania
- Slovakia (2):
  - Jesenius Faculty of Medicine in Martin, Clinic of Gastroenterological Internal Medicine, Slovak Republic, Martin
  - Department of Internal Medicine, University Hospital Trnava, Slovak Republic, Trnava
- Department of Surgical Gastroenterology, Karolinska University Hospital, Stockholm, Sweden, Stockholm, Sweden
- King's Institute of Therapeutic Endoscopy, London, UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martinek J, Hustak R, Mares J, Vackova Z, Spicak J, Kieslichova E, Buncova M, Pohl D, Amin S, Tack J. Endoscopic pyloromyotomy for the treatment of severe and refractory gastroparesis: a pilot, randomised, sham-controlled trial. Gut. 2022 Nov;71(11):2170-2178. doi: 10.1136/gutjnl-2022-326904. Epub 2022 Apr 25. PMID 35470243